CLINICAL TRIAL: NCT03268499
Title: Ethiodized Oil-based Transarterial Chemoembolization for Patients With Hepatocellular Carcinoma: A Randomized Controlled Trial of Aqueous Cisplatin Emulsion Versus Anhydrous Cisplatin Suspension
Brief Title: Emulsion Versus Suspension in Chemoembolization for Hepatocellular Carcinoma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Simon Yu, Professor, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: VIR-14-07
Record Dates: First submitted 2017-08-29; First posted 2017-08-31 (Actual); Results first posted 2024-11-15 (Actual); Last update posted 2024-11-15 (Actual); Status verified 2024-03

CONDITIONS: Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Intervention Model Description: prospective, multi-center, parallel-group, open-label, phase III randomized control trial
Who Masked: Investigator, Outcomes Assessor
Masking Description: The patients, doctors and other caretakers are not blinded to group allocation. Data collectors and analysts who assessed the study outcome and radiologists who assessed tumor response are blinded to group allocation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Suspension Group (Experimental): Patients are treated with chemoembolization using a formulation that consists of a suspension of 100mg pure anhydrous cisplatin in 20mL Lipiodol (5mg cisplatin /mL suspension)
  Interventions: Procedure: Lipiodol-based transarterial chemoembolization
- Emulsion Group (Active Comparator): Patients are treated with chemoembolization using a formulation that consists of 10mg aqueous cisplatin (10mL) mixed with 10mL Lipiodol to form an emulsion (0.5mg cisplatin/mL emulsion)
  Interventions: Procedure: Lipiodol-based transarterial chemoembolization

INTERVENTIONS:
Procedure: Lipiodol-based transarterial chemoembolization — Arterial catheterization to segmental, subsegmental, or sub-subsegmental level was achieved depending on the tumor size, to gain arterial access as close to the tumors as possible. The formulation was delivered under fluoroscopic control until the vasculature of all tumors was entirely filled, or until the maximum dose was reached.
  Other Names: Conventional chemoembolization; cTACE

SUMMARY:
The aim of the study was to evaluate the safety and efficacy of using the new formulation (Lipiodol-cisplatin suspension) for TACE in the treatment of HCC as compared to the conventional formulation (Lipiodol-cisplatin emulsion). This is a prospective, parallel-group, open-label randomized, phase III study that is conducted in accordance to the Declaration of Helsinki and international standards of Good Clinical Practice, and approved by the institutional review board. Eligible patients were randomized into either a treatment arm of Lipiodol-cisplatin suspension or a control arm of Lipiodol-cisplatin emulsion with a 1:1 ratio.

DETAILED DESCRIPTION:
Randomization with 1:1 ratio is centralized and performed by an independent statistician, it is stratified by the diameter of largest tumor less than or equal to 5cm or > 5cm, and total number of tumors less than or equal to 3 or > 3. Random permuted block method with block size of 4 to 6 is used according to a computer-generated allocation sequence. The patients, doctors and other caretakers are not blinded to group allocation. Data collectors and analysts who assess the study outcome and radiologists who assess tumor response are blinded to group allocation.

Assuming the complete response rates in the Suspension Group and Emulsion Group are 70% and 35% respectively, 85% power and 5% level of confidence, the sample size is estimated to be 70 (35 for each arm). Assuming 10 subjects to be withdrawn from the study or lost to follow-up, the final sample size is estimated to be 80.

ELIGIBILITY:
Inclusion criteria

1. Written informed consent
2. Age above 18 years
3. HCC unsuitable for resection or ablation
4. Child-Pugh A cirrhosis
5. Eastern Cooperative Oncology Group performance score 0 or 1
6. BCLC A or B
7. No previous treatment for HCC except for liver resection
8. HCC diagnosed by typical enhancement patterns on cross sectional imaging or histology.
9. No extra-hepatic involvement on non-enhanced CT thorax and triphasic contrast enhanced CT abdomen.
10. No invasion of portal vein or hepatic vein
11. Massive expansive tumor morphology with measurable lesion on CT (characterized by well-defined spherical or globular configuration, with or without tumor capsule or satellite lesions)
12. Total tumor mass < 50% liver volume
13. Size of any individual tumor greater than or equal to 10cm in largest dimension
14. Serum creatinine < 130 umol/L or Creatinine clearance > 55 ml/min.

Exclusion criteria

1. Known active malignancy within the last 3 years
2. History of acute tumor rupture presenting with hemo-peritoneum
3. Biliary obstruction not amenable to percutaneous or endoscopic drainage
4. History of hepatic encephalopathy
5. Intractable ascites not controllable by medical therapy
6. History of variceal bleeding within last 3 months
7. Infiltrative tumor morphology (characterized by ill- defined tumor margin and amorphous configuration) or diffuse tumor morphology (characterized by large number of small nodules)
8. Un-correctable Arterio-portal venous shunt affecting >1 hepatic segment on CT
9. Arterial-hepatic venous shunt with hepatic vein opacified in arterial phase on CT

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2016-09-09 (Actual); Primary Completion 2023-02-28 (Actual); Study Completion 2023-04-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Simon Yu, Principal Investigator — DIIR, CUHK, Hong Kong
Locations (1):
- Department of Imaging and Interventional Radiology, Prince of Wales Hospital, The Chinese University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Yu SCH, Chan L, Lee KF, Cho CCM, Hui EP, Chu CCM, Cheung SYS, Lok HT, Li L, Wong JKT, Wong JC, Yuen TY, Yu PSM, Wong SSM, Wong HL, Ho CHCH, Mo F, Yeo WMM. Ethiodized Oil-based Transarterial Chemoembolization for Hepatocellular Carcinoma: Randomized Clinical Trial of Anhydrous Cisplatin Suspension versus Cisplatin Emulsion. Radiology. 2025 Nov;317(2):e242982. doi: 10.1148/radiol.242982. PMID 41288481

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment period: September 2016 to August 2022
  Recruitment took place in the surgery and oncology clinics of three general hospitals including Prince of Wales Hospital, United Christian Hospital and Tuen Mun Hospital in Hong Kong
Pre-assignment Details: Of all 2772 new HCC patients who attended the three hospitals from September 2016 to August 2022, 862 patients who refused or were considered unsuitable for liver resection or ablation were screened, 782 patients were excluded due to failing to meet the eligibility criteria (97%) or having declined to participate (3%).
Period: Overall Study
Arm/Group | Emulsion Group | Suspension Group
Started | 40 | 40
Completed | 38 (2 patients did not receive treatment because these patients withdrew themselves from the study) | 39 (1 patient did not receive treatment because this patient withdrew himself from the study)
Not Completed | 2 | 1
Not completed — Withdrawal by Subject | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Suspension Group: Received TACE using suspension formulation
- Emulsion Group: Received TACE using emulsion formulation
- Total: Total of all reporting groups
Arm/Group | Suspension Group | Emulsion Group | Total
Number analyzed (Participants) | 39 | 38 | 77
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 13 | 14 | 27
  >=65 years | 26 | 24 | 50
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 70 [64 to 75] | 68 [62.8 to 72.8] | 68 [64 to 75]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 5 | 18
  Male | 26 | 33 | 59
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 39 | 38 | 77
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Hong Kong | 39 | 38 | 77

OUTCOME MEASURES:

1. Primary Outcome: Number of Paticipants With Complete Tumor Response After the First 3 Treatments
Description: Complete tumor response is defined according to the Modified Response Evaluation Criteria in Solid Tumors (mRECIST) criteria as well as DSA findings during the second and third treatment, it is defined as the absence of enhancing tumor on CT and/ or absence of residual tumor on selective DSA of the feeding arteries to the tumors and absence of enhancing tumor on the subsequent CT.
Time Frame: Within 6 months after randomization
Measure: Count of Participants; unit: Participants
Groups:
- Suspension Group; Emulsion Group: complete tumor response after the first 3 treatments
Arm/Group | Suspension Group | Emulsion Group
Number analyzed (Participants) | 39 | 38
Participants | 35 | 18

2. Primary Outcome: Number of Participants With Severe Adverse Events of All Treatment Procedures Occurring Within 30 Days of the Treatment
Description: Severe adverse events is defined as any undesirable symptom, sign or medical condition which was fatal or life-threatening, required or prolonged hospitalization, resulted in persistent or significant disability/incapacity, or was medically significant, might jeopardize the patient and might require medical or surgical intervention.
Time Frame: within 30 days of the treatment
Measure: Count of Participants; unit: Participants
Groups:
- Suspension Group; Emulsion Group: Incidence of serious adverse event within 30 days of all treatments
Arm/Group | Suspension Group | Emulsion Group
Number analyzed (Participants) | 39 | 38
Participants | 2 | 7

3. Secondary Outcome: Number of Paticipants With Complete Tumour Response After the First Treatment
Description: as for outcome 1
Time Frame: At 3 months after the first treatment
Measure: Count of Participants; unit: Participants
Groups:
- Suspension Group; Emulsion Group: Complete response after the first treatment
Arm/Group | Suspension Group | Emulsion Group
Number analyzed (Participants) | 39 | 38
Participants | 22 | 4

4. Secondary Outcome: Number of Participants With Complete or Partial Tumour Response at 6 Months
Description: Objective tumor response was defined as complete response or partial response. Partial response was defined by the modified RECIST criteria as at least a 30% decrease in the sum of diameters of viable (enhancement in the arterial phase) target lesions, taking as reference the baseline sum of the diameters of target lesions
Time Frame: At 6 months after the first treatment
Measure: Count of Participants; unit: Participants
Groups:
- Suspension Group; Emulsion Group: Objective tumor response in first 6 months
Arm/Group | Suspension Group | Emulsion Group
Number analyzed (Participants) | 39 | 38
Participants | 39 | 27

5. Secondary Outcome: Number of Participants With Intralesional Tumour Progression From Randomization Date up to 78 Months
Description: Intralesional tumor progression is defined as tumor recurrence at the site of treated tumor after initial complete tumor response, or any degree of enlargement of treated tumor after initial partial response;
Time Frame: throughout follow-up period, up to 78 months
Population: 2 participants excluded from analysis in each group since the patients received liver resection
Measure: Count of Participants; unit: Participants
Groups:
- Suspension Group; Emulsion Group: Intralesional tumor progression throughout follow up period
Arm/Group | Suspension Group | Emulsion Group
Number analyzed (Participants) | 37 | 36
Participants | 5 | 17

6. Secondary Outcome: Number of Participants With Extralesional Tumour Progression From Randomization Date up to 78 Months
Description: Extralesional tumor progression is defined as occurrence of new tumor at a new site of the liver;
Time Frame: throughout follow-up period, up to 78 months
Measure: Count of Participants; unit: Participants
Groups:
- Suspension Group; Emulsion Group: Extralesional tumour progression
Arm/Group | Suspension Group | Emulsion Group
Number analyzed (Participants) | 37 | 36
Participants | 12 | 20

7. Secondary Outcome: Number of Participants With Extrahepatic Tumour Progression up to 78 Months
Description: Extrahepatic tumor progression is defined as occurrence of venous invasion by tumor or extrahepatic tumor metastasis;
Time Frame: throughout follow-up period, up to 78 months
Measure: Count of Participants; unit: Participants
Groups:
- Suspension Group; Emulsion Group: Extrahepatic progression
Arm/Group | Suspension Group | Emulsion Group
Number analyzed (Participants) | 37 | 36
Participants | 3 | 3

8. Secondary Outcome: Time Interval in Months From Randomization Date to Occurrence of Any Kind of Tumor Progression up to 78 Months
Description: Any kind of tumor progression include intralesional progression, extralesional progression, or extrahepatic progression
Time Frame: throughout follow-up period, up to 78 months
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Suspension Group; Emulsion Group: Time to any kind of tumor progression
Arm/Group | Suspension Group | Emulsion Group
Number analyzed (Participants) | 37 | 36
months | 24.6 [13.3 to 38.9] | 10.7 [7.5 to 14.1]

9. Secondary Outcome: Progression Free Survival in Number of Months up to 78 Months
Description: Progression free survival is defined as the interval between the randomization date and the date of any kind of tumor progression or death from any cause;
Time Frame: throughout follow-up period, up to 78 months
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Suspension Group; Emulsion Group: Progression free survival
Arm/Group | Suspension Group | Emulsion Group
Number analyzed (Participants) | 37 | 36
months | 21.1 [14.3 to 38.9] | 10.4 [7.3 to 13.4]

10. Secondary Outcome: Overall Survival in Months up to 78 Months
Description: Overall survival Overall survival is defined as the interval between the randomization date and the date of death from any cause. In the absence of confirmation of death, survival time was censored at the last date the patient was known to be alive;
Time Frame: throughout follow-up period, up to 78 months
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Suspension Group; Emulsion Group: Overall survival
Arm/Group | Suspension Group | Emulsion Group
Number analyzed (Participants) | 37 | 36
months | 53.3 [40.5 to 80] | 36 [25.7 to 46.6]

11. Secondary Outcome: Adverse Event
Description: Number of participants with the specific adverse event that occurred within 30 days after the first treatment
Time Frame: Within 30 days after the first treatment
Measure: Count of Participants; unit: Participants
Groups:
- Suspension Group; Emulsion Group: Adverse event
Arm/Group | Suspension Group | Emulsion Group
Number analyzed (Participants) | 39 | 38
Participants
  Fever | 30 | 32
  Nausea | 14 | 8
  Vomiting | 13 | 10
  Abdominal pain | 25 | 26
  bilirubin elevation | 32 | 37
  albumin depression | 33 | 30
  Alkaline phosphatase elevation | 31 | 33
  Alanine aminotransferase | 39 | 33

12. Secondary Outcome: Serious Adverse Event
Description: Serious adverse event that occurs within 30 days after all treatments
Time Frame: Within 30 days after all treatments
Measure: Count of Participants; unit: Participants
Groups:
- Suspension; Emulsion: Serious adverse event
Arm/Group | Suspension | Emulsion
Number analyzed (Participants) | 39 | 38
Participants | 2 | 7

ADVERSE EVENTS:
Time Frame: Up to 78 months after randomization
Description: Details of "Adverse events" are being reported under secondary endpoints. "All-cause mortality", details of "Serious Adverse Events", and "Other Adverse Events" are being reported here.
Groups:
- Suspension Group; Emulsion Group: Details are provided under "Adverse events" in secondary endpoints.
Arm/Group | Suspension Group | Emulsion Group
All-Cause Mortality (participants affected / at risk) | 10/39 | 16/38
Serious Adverse Events (participants affected / at risk) | 2/39 | 7/38
Other Adverse Events (participants affected / at risk) | 39/39 | 38/38
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Suspension Group (N=39) | Emulsion Group (N=38)
Death (Hepatobiliary disorders) | 0 (0) | 1 (1) — death
Liver abscess (Hepatobiliary disorders) | 1 (1) | 4 (4)
Biliary sepsis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Bleeding varices (Gastrointestinal disorders) | 0 (0) | 1 (1)
Liver failure (Hepatobiliary disorders) | 1 (1) | 1 (1)
Gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Suspension Group (N=39) | Emulsion Group (N=38)
Fever (General disorders) | 30 (30) | 32 (32)
Nausea (General disorders) | 14 (14) | 8 (8)
Vomiting (General disorders) | 13 (13) | 10 (10)
Abdominal pain (Hepatobiliary disorders) | 25 (25) | 26 (26)
Bilirubin elevation (Hepatobiliary disorders) | 32 (32) | 37 (37)
Albumin depression (Hepatobiliary disorders) | 33 (33) | 30 (30)
Alkaline phosphatase elevation (Hepatobiliary disorders) | 31 (31) | 33 (33)
Alanine aminotransferase elevation (Hepatobiliary disorders) | 39 (39) | 33 (33)

LIMITATIONS AND CAVEATS:
The number of subjects was relatively small, although the power of study was 85%. Using CT in assessing tumor response in the presence of intratumoral ethiodized oil may suffer a higher risk of missing minute tumors hidden among the ethiodized oil cast and over-diagnosing complete tumor response, however, the study outcomes were unlikely significantly affected, because viable tumors that were missed would have been captured at the study endpoint of intralesional tumor progression.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2016-07-16): https://cdn.clinicaltrials.gov/large-docs/99/NCT03268499/Prot_000.pdf
  • Statistical Analysis Plan (2016-07-16): https://cdn.clinicaltrials.gov/large-docs/99/NCT03268499/SAP_001.pdf
  • Informed Consent Form (2016-07-16): https://cdn.clinicaltrials.gov/large-docs/99/NCT03268499/ICF_002.pdf